CLINICAL TRIAL: NCT04270006
Title: Effect of Adipose Derived Stem Cells Exosomes as an Adjunctive Therapy to Scaling and Root Planning in the Treatment of Periodontitis: A Human Clinical Trial
Brief Title: Evaluation of Adipose Derived Stem Cells Exo.in Treatment of Periodontitis
Acronym: exosomes
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ebtehal Mohammed, Lecturer of oral medicine, periodontotlogy and oral diagnosis, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDBSUREC/21012020/ME
Record Dates: First submitted 2020-02-08; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Periodontitis
Keywords: Periodontitis; SRP; ADSCs; Exosomes; treatment
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exosomes (Experimental)
  Interventions: Biological: adipose derived stem cells exosomes

INTERVENTIONS:
Biological: adipose derived stem cells exosomes — they are small extracellular vesicles

SUMMARY:
The adipose stem cells exosomes will be extracted from adipose stem cells isolated autogenously from the patient to be injected locally into the periodontal pockets in order to evaluate their regenerative effect.

ELIGIBILITY:
Inclusion Criteria:

* Advanced periodontitis (Stage III or IV)
* Healthy patients.

Exclusion Criteria:

* Smokers, Diabetic, Pregnant ladies, Under corticosteroids or contraceptive treatment,poor oral hygiene.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-09-12 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
change in gingival inflammation | 0, 3 and 6 months
  Gingival index (GI)
change in pocket depth | 0, 3 and 6 months
  Probing depth (PD)
change in attachment level | 0, 3 and 6 months
  Clinical attachment level (CAL)
change in Bone level | 0 and 6 months
  Cone beam C.T (CBCT)

CONTACTS AND LOCATIONS:
Overall Officials: Ebtehal Mohammed, Ph.D, Principal Investigator — Lecturer of Oral Medicine , Oral diagnosis and Periodontology , Faculty of Dentistry, Beni- Suef University.; Nesrine Mohammed Khairy, Associated Professor, Study Director — Oral and Maxillofacial Surgery, Faculty of Dentistry, Cairo University; Noha Saleh Mohammed, Associated, Study Director — Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University.; Dina Sabry, Professor, Study Director — Biochemistry, Faculty of Medicine, Cairo University
Locations (2):
- Egypt (2):
  - Beni-Suef University, Banī Suwayf
  - Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: Yes
the data will be published
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: the data will be available after at least one year